CLINICAL TRIAL: NCT03885076
Title: Assessing Feasibility of Expansion and Characterization of Gamma Delta T Cells From Peripheral Blood and Bone Marrow of Patients With Acute Myeloid Leukaemia as Starting Product for Generation of CD33-CD28 Gamma Delta T Cells
Brief Title: Gamma Delta T Cells in AML
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Royal Marsden NHS Foundation Trust (Other)
Collaborators: TC Biopharm (Industry)
Responsible Party: Sponsor
Other Study IDs: CCR4877
Record Dates: First submitted 2019-03-20; First posted 2019-03-21 (Actual); Last update posted 2019-07-02 (Actual); Status verified 2019-06

CONDITIONS: Acute Myeloid Leukemia
MeSH Terms: conditions — Leukemia, Myeloid, Acute

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Acute myeloid leukaemia: Patients with Acute Myeloid Leukaemia (excluding M3) at presentation, remission or with refractory or relapsed disease. There is no intervention. This is an observational tissue collection study.
  Interventions: Procedure: Blood collection and bone marrow aspirate

INTERVENTIONS:
Procedure: Blood collection and bone marrow aspirate — Blood and bone marrow samples will be collected for the trial alongside routine tests.

SUMMARY:
The Royal Marsden NHS Foundation Trust is committed to improving patient experience; this research is being undertaken to try to develop a novel treatment for patients with Acute Myeloid Leukaemia (AML). Researchers aim to develop a new therapy which uses a patient's own immune cells called T cells to treat AML. In this study, numbers and properties of T cells which can be collected from the blood of patients with AML at various points throughout their treatment will be investigated. Blood samples will be collected at the same time as the patient's bone marrow test.

If patients need further bone marrow tests during their course of treatment to assess the status of disease, the research team would ask that additional samples are taken at the same time as the bone marrow and blood will be collected at the same time as the routine blood draw.

Following collection of blood samples, they will be used to purify a population of blood cells called Gamma Delta T cells which have been shown to have a potential role in control of cancers. In addition the researchers plan to determine whether it is possible to put a novel receptor called a chimeric antigen receptor (CAR) to potentially directly target leukaemia cells. Currently this is only an exploratory study and none of the samples collected will be used for treatment and is only to assess whether or not this strategy is feasible. This may however lead on to studies in the future looking at the safety and effectiveness of this strategy. This hopefully will lead in the future to improvements in treatment and outcome for patients with AML.

If patients need further bone marrow tests during their course of treatment to assess the status of disease, the research team would ask that additional samples are taken at the same time as the bone marrow and blood will be collected at the same time as the routine blood draw.

Following collection of blood samples, they will be used to purify a population of blood cells called Gamma Delta T cells which have been shown to have a potential role in control of cancers. In addition the researchers plan to determine whether it is possible to put a novel receptor called a chimeric antigen receptor (CAR) to potentially directly target leukaemia cells. Currently this is only an exploratory study and none of the samples collected will be used for treatment and is only to assess whether or not this strategy is feasible. This may however lead on to studies in the future looking at the safety and effectiveness of this strategy. This hopefully will lead in the future to improvements in treatment and outcome for patients with AML.

ELIGIBILITY:
Inclusion Criteria:

1. Patients over the age of 18 at time of diagnosis or at time of relapse of disease
2. Patients with Acute Myeloid Leukaemia (excluding M3) at presentation, remission or with refractory or relapsed disease.
3. Patients must have given informed written consent to participate in this study.

Exclusion Criteria:

1. Uncontrolled systemic infection
2. Currently receiving corticosteroids or other immune-suppressants treatment (except in cases where the patient is receiving treatment with replacement doses for adrenal insufficiency)
3. Treatment with bisphosphonates, for instance zoledronate, in the previous 3 months or throughout the trial
4. Active, known or suspected autoimmune disease such as Ulcerative Colitis / Inflammatory bowel disease, Addison's disease
5. Pregnancy or lactation before or during the study
6. Substance abuse, medical, psychological or social conditions that may interfere with the subject's participation in the study
7. Patients with active Hepatitis B, C or HIV will be excluded from this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with newly diagnosed AML or relapsed/refractory AML
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2018-08-23 (Actual); Primary Completion 2020-03 (Estimated); Study Completion 2021-03 (Estimated)

PRIMARY OUTCOMES:
Percentage viable gamma delta T cells | 6 months
  % of viable Vd2g T cells that can be generated from peripheral blood and bone marrow samples from AML patients at diagnosis and in AML patients with relapsed/refractory disease

SECONDARY OUTCOMES:
Transduced cells | 6 months
  % of Vd2g T cells transduced with a CAR.
Target AML cells killed | 6 months
  % of target AML cells killed by Gamma Delta CAR-T cells
Target monocytes killed | 6 months
  % of target monocytes killed by Gamma Delta Car T cells

CONTACTS AND LOCATIONS:
Overall Officials: Emma Nicholson, Principal Investigator — Royal Marsden NHS Foundation Trust
Locations (1):
- The Royal Marsden NHS Foundation Trust, Sutton, United Kingdom

IPD SHARING:
Plan to Share IPD: No